CLINICAL TRIAL: NCT01150045
Title: A Phase III Trial of 6 Versus 12 Treatments of Adjuvant FOLFOX Plus Celecoxib or Placebo for Patients With Resected Stage III Colon Cancer
Brief Title: Oxaliplatin, Leucovorin Calcium, and Fluorouracil With or Without Celecoxib in Treating Patients With Stage III Colon Cancer Previously Treated With Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CALGB-80702; U10CA031946 (NIH); CALGB-80702; CDR0000675693 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2010-06-23; First posted 2010-06-24 (Estimated); Results first posted 2021-08-06 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; stage III colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Celecoxib; Fluorouracil; Oxaliplatin; Leucovorin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A - FOLFOX and placebo (12 treatments) (Active Comparator): Patients receive FOLFOX every 2 weeks plus placebo every day for 12 treatments (24 weeks). Each 2-week period is called a cycle. FOLFOX includes oxaliplatin, leucovorin and 5-FU.Then, patients receive placebo alone every day for 3 years total.
  Interventions: Drug: 5-fluorouracil; Other: placebo; Drug: oxaliplatin; Drug: leucovorin
- Arm B - FOLFOX and celecoxib (12 treatments) (Experimental): Patients receive FOLFOX every 2 weeks plus celecoxib every day for 12 treatments (24 weeks). Each 2-week period is called a cycle. FOLFOX includes oxaliplatin, leucovorin and 5-FU.Then, patients receive celecoxib alone every day for 3 years total.
  Interventions: Drug: celecoxib; Drug: 5-fluorouracil; Drug: oxaliplatin; Drug: leucovorin
- Arm C - FOLFOX and placebo (6 treatments) (Active Comparator): Patients receive FOLFOX every 2 weeks plus placebo every day for 6 treatments (12 weeks). Each 2-week period is called a cycle. FOLFOX includes oxaliplatin, leucovorin and 5-FU.Then, patients receive placebo alone every day for 3 years total.
  Interventions: Drug: 5-fluorouracil; Other: placebo; Drug: oxaliplatin; Drug: leucovorin
- Arm D - FOLFOX and celecoxib (6 treatments) (Experimental): Patients receive FOLFOX every 2 weeks plus celecoxib every day for 6 treatments (12 weeks). Each 2-week period is called a cycle. FOLFOX includes oxaliplatin, leucovorin and 5-FU.Then, patients receive celecoxib alone every day for 3 years total.
  Interventions: Drug: celecoxib; Drug: 5-fluorouracil; Drug: oxaliplatin; Drug: leucovorin

INTERVENTIONS:
Drug: celecoxib — Patients receive celecoxib 400 mg administered by mouth, once daily.
  Arms: Arm B - FOLFOX and celecoxib (12 treatments); Arm D - FOLFOX and celecoxib (6 treatments)
Drug: 5-fluorouracil — Patients receive 400 mg/m^2 intravenous bolus then 2400 mg/m^2 continuous intravenous infusion over 46-48 hours.
Other: placebo — Patients receive placebo administered by mouth, once daily.
  Arms: Arm A - FOLFOX and placebo (12 treatments); Arm C - FOLFOX and placebo (6 treatments)
Drug: oxaliplatin — Patients receive 85 mg/m^2 intravenous over two hours.
Drug: leucovorin — Patients receive 400 mg/m^2 intravenous over two hours.

SUMMARY:
PURPOSE: This randomized phase III trial is studying giving oxaliplatin, leucovorin calcium, and fluorouracil together to compare how well they work when given together with or without celecoxib in treating patients with stage III colon cancer previously treated with surgery.

RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, leucovorin calcium, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether giving oxaliplatin, leucovorin calcium, and fluorouracil is more effective with or without celecoxib in treating colon cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a multicenter study. Patients are stratified according to number of positive lymph nodes* (1-3 vs 4 or more) and concurrent regular low-dose of aspirin (yes vs no). Patients are randomized to 1 of 4 treatment arms. Please see the "Arms" section for more information. In all arms, treatment with celecoxib or placebo continues for 3 years in the absence of disease progression or unacceptable toxicity. Blood and tissue samples maybe collected for biomarker analysis and pharmacogenomic studies. The primary and secondary objectives for the research study are described below.

Primary objective:

1. To compare disease-free survival of patients with stage III colon cancer randomized to standard chemotherapy only FOLFOX or standard chemotherapy FOLFOX with 3 years of celecoxib 400 mg daily.

Secondary objectives:

1. To contribute to an international prospective pooled analysis that will compare disease-free survival of patients with stage III colon cancer randomized to 6 treatments of adjuvant FOLFOX chemotherapy or 12 treatments of adjuvant FOLFOX chemotherapy.
2. To compare overall survival of patients with stage III colon cancer randomized to standard chemotherapy only (FOLFOX) or standard chemotherapy (FOLFOX) with 3 years of celecoxib 400 mg daily.
3. To contribute to an international prospective pooled analysis that will compare overall survival of patients with stage III colon cancer randomized to 6 treatments of adjuvant FOLFOX chemotherapy or 12 treatments of adjuvant FOLFOX chemotherapy or 12 treatments of adjuvant FOLFOX chemotherapy.
4. To assess toxicities of celecoxib as maintenance adjuvant therapy in patients with stage III colon cancer.
5. To assess differences in cardiovascular-specific events with celecoxib versus placebo in a population of stage III colon cancer survivors.
6. To evaluate differences in toxicities, particularly cumulative peripheral neuropathy, for patients treated with 6 treatments of FOLFOX compared to those treated with 12 treatments of FOLFOX.

After completion of study therapy, patients are followed up every 6 months for up to 6 years.

ELIGIBILITY:
1. Requirements for tumor parameters

   1. Histologically documented adenocarcinoma of the colon. The gross inferior (caudad) margin of the primary tumor must lie above the peritoneal reflection (i.e., patients with rectal cancer are not eligible). Surgeon confirmation that the entire tumor was above the peritoneal reflection is only required in cases where it is important to establish if the tumor is a rectal or colon primary.
   2. Tumors must have been completely resected. In patients with tumor adherent to adjacent structures, en bloc R0 resection must be documented in the operative report or otherwise confirmed by the surgeon. Near or positive radial margin are not exclusions as long as en bloc resection was performed. Positive proximal margin or distal margin is an exclusion.
   3. Node positive disease (N1 or N2) as designated in AJCC version 7. Either at least one pathologically confirmed positive lymph node or N1C (defined as tumor deposit(s) in the subserosa, mesentery, or nonperitonealized pericolic or perirectal tissues without regional lymph node metastases). Patients with resected stage IV disease are not eligible.
   4. No evidence of residual involved lymph node disease or metastatic disease at the time of registration.
   5. Patients with synchronous colon cancers are eligible and staging for stratification will be based on higher N stage of the more advanced primary tumor. However, patients with synchronous colon and rectal primary tumors are not eligible.
2. NSAID use

   Patients are ineligible if they plan on regular use of NSAIDs at any dose more than 2 times per week (on average) or aspirin at more than 325 mg at least three times per week, on average. Low-dose aspirin not exceeding 100 mg/day is permitted. Patients who agree to stop regular NSAIDs or higher dose aspirin are eligible and no was out period is required.
3. Patient history

   1. No previous or concurrent malignancy, except treated basal cell or squamous cell cancer of skin, treated in situ cervical cancer, treated lobular or ductal carcinoma in situ in one breast, or any other cancer for which the patient has been disease-free for at least 5 years.
   2. No neurosensory or neuromotor toxicity ≥ grade 2 at the time of registration.
   3. No known allergy to platinum compounds.
   4. No prior allergic reaction or hypersensitivity to sulfonamides, celecoxib or NSAIDs.
   5. No history of upper gastrointestinal ulceration, upper gastrointestinal bleeding, or upper gastrointestinal perforation within the past 3 years. Patients with ulceration, bleeding or perforation in the lower bowel are not excluded.
   6. No symptomatic pulmonary fibrosis or interstitial pneumonitis ≥ grade 2.
   7. No cardiac risk factors including:

      * Uncontrolled high blood pressure (systolic blood pressure > 150).
      * Unstable angina.
      * History of documented myocardial infarction or cerebrovascular accident.
      * New York Heart Association class III or IV heart failure.
4. Pregancy/nursing status

   Non-pregnant and not nursing. Men and women of childbearing potential must agree to employ adequate contraception for the duration of chemotherapy and for as many as 8 weeks after the completion of chemotherapy due to the unknown teratogenic effects of FOLFOX on the developing fetus.
5. Age and performance status

   1. ECOG performance status 0, 1 or 2.
   2. Age at least 18 years.
6. Required initial laboratory values

   1. Granulocytes ≥ 1,500/μL
   2. Platelet count ≥ 100,000/μL
   3. Creatinine ≤ 1.5 times upper limit of normal (ULN)
   4. Total Bilirubin ≤ 1.5 times ULN in the absence of Gilbert's disease
   5. Direct bilirubin ≤ 1.5 x upper limit of normal for patients with Gilbert's syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2527 (Actual)
Dates: Start 2010-06; Primary Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Meyerhardt, MD, MPH, Study Chair — Dana-Farber Cancer Institute
Locations (842):
- United States (826):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center-Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Hospitals, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - John Muir Medical Center-Concord, Concord, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, California
  - University Oncology Associates, Fresno, California
  - California Cancer Center - North Fresno, Fresno, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Marin General Hospital, Greenbrae, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health-Chao Family Comprehensive Cancer Center, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Stanford Cancer Institute, Palo Alto, California
  - Palchak David MD, Pismo Beach, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Salinas Valley Memorial Hospital, Salinas, California
  - Salinas Valley Memorial, Salinas, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Naval Medical Center-San Diego, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Veterans Affairs Medical Center-San Francisco, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center-Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Cancer Center-Anschutz Cancer Pavilion, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Memorial Hospital Colorado Springs, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian-Saint Lukes Medical Center-Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Sanford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - University of Florida-Gainesville, Gainesville, Florida
  - Memorial Regional Hospital-Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Robert and Carol Weissman Cancer Center at Martin Health, Stuart, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Low Country Cancer Care Associates PC, Savannah, Georgia
  - Oncare Hawaii Inc - POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Presence Saint Joseph Hospital-Chicago, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Hematology Oncology Associates -Highland Park, Highland Park, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - NorthShore Hematology Oncology-Libertyville, Libertyville, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Hematology Oncology Consultants Ltd., Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center Radiation Oncology Service at the Central Illinois Comprehensive CC, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Quincy Medical Group - Clinic, Quincy, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Cadence Cancer Center in Warrenville, Warrenville, Illinois
  - Michiana Hematology Oncology PC-Crown Point, Crown Point, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - IU Health Central Indiana Cancer Centers-Fishers, Fishers, Indiana
  - Indiana University - Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consrtium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Hematology Oncology Associates - Quad Cities, Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates - Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - JCHC McCreery Cancer Center, Fairfield, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Hays Medical Center, Hays, Kansas
  - Cancer Center of Kansas - Independence, Independence, Kansas
  - Kansas City Cancer Centers - West, Kansas City, Kansas
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas - Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Kansas City Cancer Centers - Southwest, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Stormont-Vail Regional Health Center, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas - Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Hardin Memorial Hospital, Elizabethtown, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Health Center - Covington, Covington, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - Interim LSU Public Hospital, New Orleans, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Eastern Maine Medical Center Cancer Care, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - York Hospital, York Village, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Western Maryland Regional Medical Center, Cumberland, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Kaiser Permanente - Gaithersburg Medical Center, Gaithersburg, Maryland
  - Meritus Medical Center, Hagerstown, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - MetroWest Medical Center-Framingham Union Hospital, Framingham, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional Medical Center, Milford, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Berkshire Hematology Oncology, PC, Pittsfield, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Toledo Clinic Cancer Centers - Adrian, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology-Escanaba, Escanaba, Michigan
  - Botsford Hospital, Farmington, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology-Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Lakeland Community Hospital, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon and Rectal Association, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Hematology Oncology Consultants PC-Royal Oak, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis Veterans Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center - Carrie J Babb Cancer Center, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center - Saint Peters, City of Saint Peters, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital-Joplin, Joplin, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - Kansas City Cancer Centers - South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Lakeland Hospital, Saint Joseph, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Cox Health South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute - South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Barnes-Jewish West County Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare - Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Great Plains Regional Medical Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium CCOP, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Hematology West, P.C., Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Cancer Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Henderson, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Cancer and Blood Specialists-Fort Apache, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Wentworth Douglass Hospital, Dover, New Hampshire
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center-Manchester, Manchester, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Administration New Jersey Health Care System, East Orange, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - Inspira Medical Center Woodbury, Woodbury, New Jersey
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Lovelace Medical Center at Lovelace Sandia Health System, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Elmhurst Hospital Center, Elmhurst, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Queens Hospital Center, Jamaica, New York
  - North Shore University Hospital, Manhasset, New York
  - North Shore-LIJ Health System/Center for Advanced Medicine, New Hyde Park, New York
  - Beth Israel Medical Center, New York, New York
  - Saint Luke's Roosevelt Hospital Center - Saint Luke's Division, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Faxton-Saint Luke's Healthcare, Utica, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Mountain Radiation Oncology, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Transylvania Regional Hospital, Brevard, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Angel Medical Center, Franklin, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Maria Parham Medical Center, Henderson, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Park Ridge Health, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - McDowell Hospital, Marion, North Carolina
  - Rex Cancer Center, Raleigh, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Rex Cancer Center of Wakefield, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Blue Ridge Regional Hospital, Spruce Pine, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Cleveland Clinic Cancer Center Beachwood, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel Hospital East, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Veteran Affairs Medical Center, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Oncology Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - Cleveland Clinic Foundation - Strongsville, Strongsville, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UHHS Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic - Wooster Specialty Center, Wooster, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Mercy Clinic Oklahoma Communities Inc-Norman, Norman, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - PinnacleHealth Regional Cancer Center at Polyclinic Hospital, Harrisburg, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - Geisinger Medical Oncology-Pottsville, Pottsville, Pennsylvania
  - Scranton Hematology-Oncology, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Susquehanna Cancer Center at Divine Providence Hospital, Williamsport, Pennsylvania
  - Wellspan Health - York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute - Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates, PA, Lancaster, South Carolina
  - Carolina Blood and Cancer Care, Rock Hill, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute - Spartanburg, Spartanburg, South Carolina
  - Avera Saint Luke's Hospital and Cancer Center, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Medical Associates-Oncology and Hematology, Bristol, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Tennessee Oncology PLLC- Centennial Medical Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Central Vermont Medical Center, Berlin Corners, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - White River Junction Veteran Administration Medical Center, White River Junction, Vermont
  - Medical Oncology Hematology Associates of Northern Virginia Limited, Fairfax, Virginia
  - Virginia Oncology Associates - Hampton, Hampton, Virginia
  - Memorial Hospital Of Martinsville, Martinsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Virginia Cancer Institute - West End, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Saint John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Cancer Care Northwest-Valley, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center - Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - Multicare Health System, Tacoma, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Fox Valley Hematology and Oncology, Appleton, Wisconsin
  - Aurora Cancer Care-Burlington, Burlington, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System Eau Claire Hospital-Luther Campus, Eau Claire, Wisconsin
  - Aurora Cancer Care-Southern Lakes, Elkhorn, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic - Marinette, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Aurora Advanced Healthcare Inc-Menomonee Falls, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Wheaton Franciscan Healthcare - St. Joseph, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - D N Greenwald Center, Mukwonago, Wisconsin
  - Westfields Hospital/Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Oconomowoc Memorial Hospital-ProHealth Care Inc, Oconomowoc, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic - Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic - Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (15):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Horizon Health Network-Saint John Regional Hospital, Saint John, New Brunswick
  - Cambridge Memorial Hospital, Cambridge, Ontario
  - Health Sciences North, Greater Sudbury, Ontario
  - London Regional Cancer Program, London, Ontario
  - Niagara Health System-Saint Catharines General, Saint Catharines, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - PEI Cancer Treatment Centre-Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - McGill University Department of Oncology, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- San Juan City Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Zhang GQ, Meyerhardt JA, Shi Q, Twombly T, Pederson L, Ma C, Vayrynen JP, Zhao M, Takashima Y, Shergill A, Kumar P, Couture F, Kuebler P, Krishnamurthi S, Tan B, O'Reilly EM, Giannakis M, Ogino S, Jurdi A, Sharma S, Aleshin A, Shields AF, Nowak JA. Predictive Role of Circulating Tumor DNA in Stage III Colon Cancer Treated With Celecoxib: A Post Hoc Analysis of the CALGB (Alliance)/SWOG 80702 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2025 Dec 4:e255144. doi: 10.1001/jamaoncol.2025.5144. Online ahead of print. PMID 41343176
- [Derived] Nowak JA, Twombly T, Ma C, Shi Q, Haruki K, Fujiyoshi K, Vayrynen J, Zhao M, Knight J, Mane S, Shergill A, Kumar P, Couture F, Kuebler P, Krishnamurthi S, Tan B, Philip P, O'Reilly EM, Shields AF, Ogino S, Fuchs CS, Meyerhardt JA. Improved Survival With Adjuvant Cyclooxygenase 2 Inhibition in PIK3CA-Activated Stage III Colon Cancer: CALGB/SWOG 80702 (Alliance). J Clin Oncol. 2024 Aug 20;42(24):2853-2859. doi: 10.1200/JCO.23.01680. Epub 2024 Jun 18. PMID 38889377
- [Derived] Lee S, Ma C, Shi Q, Meyers J, Kumar P, Couture F, Kuebler P, Krishnamurthi S, Lewis D, Tan B, O'Reilly EM, Shields AF, Meyerhardt JA. Sleep and cancer recurrence and survival in patients with resected Stage III colon cancer: findings from CALGB/SWOG 80702 (Alliance). Br J Cancer. 2023 Aug;129(2):283-290. doi: 10.1038/s41416-023-02290-2. Epub 2023 May 13. PMID 37179438
- [Derived] Cheng E, Shi Q, Shields AF, Nixon AB, Shergill AP, Ma C, Guthrie KA, Couture F, Kuebler P, Kumar P, Tan B, Krishnamurthi SS, Ng K, O'Reilly EM, Brown JC, Philip PA, Caan BJ, Cespedes Feliciano EM, Meyerhardt JA. Association of Inflammatory Biomarkers With Survival Among Patients With Stage III Colon Cancer. JAMA Oncol. 2023 Mar 1;9(3):404-413. doi: 10.1001/jamaoncol.2022.6911. PMID 36701146
- [Derived] Lee S, Ma C, Shi Q, Kumar P, Couture F, Kuebler P, Krishnamurthi S, Lewis D, Tan B, Goldberg RM, Venook A, Blanke C, O'Reilly EM, Shields AF, Meyerhardt JA. Potential Mediators of Oxaliplatin-Induced Peripheral Neuropathy From Adjuvant Therapy in Stage III Colon Cancer: Findings From CALGB (Alliance)/SWOG 80702. J Clin Oncol. 2023 Feb 10;41(5):1079-1091. doi: 10.1200/JCO.22.01637. Epub 2022 Nov 11. PMID 36367997
- [Derived] Gallois C, Shi Q, Meyers JP, Iveson T, Alberts SR, de Gramont A, Sobrero AF, Haller DG, Oki E, Shields AF, Goldberg RM, Kerr R, Lonardi S, Yothers G, Kelly C, Boukovinas I, Labianca R, Sinicrope FA, Souglakos I, Yoshino T, Meyerhardt JA, Andre T, Papamichael D, Taieb J. Prognostic Impact of Early Treatment and Oxaliplatin Discontinuation in Patients With Stage III Colon Cancer: An ACCENT/IDEA Pooled Analysis of 11 Adjuvant Trials. J Clin Oncol. 2023 Feb 1;41(4):803-815. doi: 10.1200/JCO.21.02726. Epub 2022 Oct 28. PMID 36306483
- [Derived] Meyerhardt JA, Shi Q, Fuchs CS, Meyer J, Niedzwiecki D, Zemla T, Kumthekar P, Guthrie KA, Couture F, Kuebler P, Bendell JC, Kumar P, Lewis D, Tan B, Bertagnolli M, Grothey A, Hochster HS, Goldberg RM, Venook A, Blanke C, O'Reilly EM, Shields AF. Effect of Celecoxib vs Placebo Added to Standard Adjuvant Therapy on Disease-Free Survival Among Patients With Stage III Colon Cancer: The CALGB/SWOG 80702 (Alliance) Randomized Clinical Trial. JAMA. 2021 Apr 6;325(13):1277-1286. doi: 10.1001/jama.2021.2454. PMID 33821899
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient withdrew from the trial before being randomized and was excluded from any analysis.
Groups:
- Arm A - 12 Cycles of FOLFOX Plus Placebo Daily: The FOLFOX regimen consisted of every 2 weeks cycles for 12 cycles of 2-hour infusions of oxaliplatin at 85 mg/m2 and leucovorin at 400 mg/m2, followed by a bolus infusion of 400-mg/m2 of fluorouracil following by 46-48-hour continuous infusion of 2400-mg/m2 of fluorouracil.
  > Placebo was dosed at 400 mg orally daily, starting by day 1 of the second treatment of FOLFOX. Placebo was administered daily for 3 years from the date of initiation of the first dose or until recurrence of disease or unacceptable toxicity.
- Arm B - 12 Cycles of FOLFOX Plus Celecoxib Daily: The FOLFOX regimen consisted of every 2 weeks cycles for 12 cycles of 2-hour infusions of oxaliplatin at 85 mg/m2 and leucovorin at 400 mg/m2, followed by a bolus infusion of 400-mg/m2 of fluorouracil following by 46-48-hour continuous infusion of 2400-mg/m2 of fluorouracil.
  > Celecoxib was dosed at 400 mg orally daily, starting by day 1 of the second treatment of FOLFOX. Celecoxib was administered daily for 3 years from the date of initiation of the first dose or until recurrence of disease or unacceptable toxicity.
- Arm C - 6 Cycles of FOLFOX Plus Placebo Daily: The FOLFOX regimen consisted of every 2 weeks cycles for 6 cycles of 2-hour infusions of oxaliplatin at 85 mg/m2 and leucovorin at 400 mg/m2, followed by a bolus infusion of 400-mg/m2 of fluorouracil following by 46-48-hour continuous infusion of 2400-mg/m2 of fluorouracil.
  > Placebo was dosed at 400 mg orally daily, starting by day 1 of the second treatment of FOLFOX. Placebo was administered daily for 3 years from the date of initiation of the first dose or until recurrence of disease or unacceptable toxicity.
- Arm D - 6 Cycles of FOLFOX Plus Celecoxib Daily: The FOLFOX regimen consisted of every 2 weeks cycles for 6 cycles of 2-hour infusions of oxaliplatin at 85 mg/m2 and leucovorin at 400 mg/m2, followed by a bolus infusion of 400-mg/m2 of fluorouracil following by 46-48-hour continuous infusion of 2400-mg/m2 of fluorouracil.
  > Celecoxib was dosed at 400 mg orally daily, starting by day 1 of the second treatment of FOLFOX. Celecoxib was administered daily for 3 years from the date of initiation of the first dose or until recurrence of disease or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A - 12 Cycles of FOLFOX Plus Placebo Daily | Arm B - 12 Cycles of FOLFOX Plus Celecoxib Daily | Arm C - 6 Cycles of FOLFOX Plus Placebo Daily | Arm D - 6 Cycles of FOLFOX Plus Celecoxib Daily
Started | 615 | 647 | 646 | 618
Completed | 615 | 646 | 646 | 617
Not Completed | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All patients that were randomized and evaluable for the primary endpoint are included in this analysis.
Groups:
- Arm A - FOLFOX and Placebo (12 Treatments): The FOLFOX regimen consisted of every 2 weeks cycles for 12 cycles of 2-hour infusions of oxaliplatin at 85 mg/m2 and leucovorin at 400 mg/m2, followed by a bolus infusion of 400-mg/m2 of fluorouracil following by 46-48-hour continuous infusion of 2400-mg/m2 of fluorouracil.> Placebo was dosed at 400 mg orally daily, starting by day 1 of the second treatment of FOLFOX. Placebo was administered daily for 3 years from the date of initiation of the first dose or until recurrence of disease or unacceptable toxicity.
- Arm B - 12 Cycles of FOLFOX Plus Celecoxib Daily: The FOLFOX regimen consisted of every 2 weeks cycles for 12 cycles of 2-hour infusions of oxaliplatin at 85 mg/m2 and leucovorin at 400 mg/m2, followed by a bolus infusion of 400-mg/m2 of fluorouracil following by 46-48-hour continuous infusion of 2400-mg/m2 of fluorouracil.> Celecoxib was dosed at 400 mg orally daily, starting by day 1 of the second treatment of FOLFOX. Celecoxib was administered daily for 3 years from the date of initiation of the first dose or until recurrence of disease or unacceptable toxicity.
- Arm C - 6 Cycles of FOLFOX Plus Placebo Daily: The FOLFOX regimen consisted of every 2 weeks cycles for 6 cycles of 2-hour infusions of oxaliplatin at 85 mg/m2 and leucovorin at 400 mg/m2, followed by a bolus infusion of 400-mg/m2 of fluorouracil following by 46-48-hour continuous infusion of 2400-mg/m2 of fluorouracil.> Placebo was dosed at 400 mg orally daily, starting by day 1 of the second treatment of FOLFOX. Placebo was administered daily for 3 years from the date of initiation of the first dose or until recurrence of disease or unacceptable toxicity.
- Arm D - 6 Cycles of FOLFOX Plus Celecoxib Daily: The FOLFOX regimen consisted of every 2 weeks cycles for 6 cycles of 2-hour infusions of oxaliplatin at 85 mg/m2 and leucovorin at 400 mg/m2, followed by a bolus infusion of 400-mg/m2 of fluorouracil following by 46-48-hour continuous infusion of 2400-mg/m2 of fluorouracil.> Celecoxib was dosed at 400 mg orally daily, starting by day 1 of the second treatment of FOLFOX. Celecoxib was administered daily for 3 years from the date of initiation of the first dose or until recurrence of disease or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Arm A - FOLFOX and Placebo (12 Treatments) | Arm B - 12 Cycles of FOLFOX Plus Celecoxib Daily | Arm C - 6 Cycles of FOLFOX Plus Placebo Daily | Arm D - 6 Cycles of FOLFOX Plus Celecoxib Daily | Total
Number analyzed (Participants) | 615 | 646 | 646 | 617 | 2524
Age, Continuous [Median (Full Range); unit: years] | 61.0 [19.3 to 86.5] | 61.9 [21.8 to 88.7] | 61.0 [20.5 to 84.4] | 61.5 [27.7 to 87.6] | 61.3 [19.3 to 88.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 265 | 297 | 296 | 276 | 1134
  Male | 350 | 349 | 350 | 341 | 1390
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 45 | 55 | 49 | 191
  Not Hispanic or Latino | 559 | 586 | 571 | 552 | 2268
  Unknown or Not Reported | 14 | 15 | 20 | 16 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 5 | 3 | 4 | 15
  Asian | 22 | 32 | 21 | 32 | 107
  Native Hawaiian or Other Pacific Islander | 0 | 4 | 2 | 1 | 7
  Black or African American | 82 | 88 | 76 | 73 | 319
  White | 487 | 500 | 522 | 488 | 1997
  More than one race | 1 | 2 | 3 | 0 | 6
  Unknown or Not Reported | 20 | 15 | 19 | 19 | 73
Region of Enrollment [Number; unit: participants]
  Canada | 57 | 44 | 70 | 61 | 232
  United States | 558 | 602 | 576 | 556 | 2292

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: Disease-Free Survival (DFS) is defined as the time of randomization until documented progression or death from any cause. The endpoint of this trial is to compare disease-free survival of patients with stage III colon cancer randomized to standard chemotherapy only (FOLFOX; Arm A and Arm C) or standard chemotherapy (FOLFOX) with 3 years of celecoxib 400 mg daily (Arm B and Arm D). The percentage of patients who were alive and disease free after 3 years are reported here. A log-rank test stratified with the stratification factors was used to compare disease-free survival (celecoxib vs placebo)
Time Frame: At 3 years of follow-up
Population: All patients that were randomized and evaluable were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- FOLFOX and Placebo (Arms A +C): Arm A
  The FOLFOX regimen consisted of every 2 weeks cycles for 12 cycles of 2-hour infusions of oxaliplatin at 85 mg/m2 and leucovorin at 400 mg/m2, followed by a bolus infusion of 400-mg/m2 of fluorouracil following by 46-48-hour continuous infusion of 2400-mg/m2 of fluorouracil.
  Placebo was dosed at 400 mg orally daily, starting by day 1 of the second treatment of FOLFOX. Placebo was administered daily for 3 years from the date of initiation of the first dose or until recurrence of disease or unacceptable toxicity.
  Arm C
  The FOLFOX regimen consisted of every 2 weeks cycles for 6 cycles of 2-hour infusions of oxaliplatin at 85 mg/m2 and leucovorin at 400 mg/m2, followed by a bolus infusion of 400-mg/m2 of fluorouracil following by 46-48-hour continuous infusion of 2400-mg/m2 of fluorouracil.
  Placebo was dosed at 400 mg orally daily, starting by day 1 of the second treatment of FOLFOX. Placebo was administered daily for 3 years from the date of initiation of the first dose or until recurrence of disease or unacceptable toxicity.
- FOLFOX Plus Celecoxib Daily (Arms B + D): Arm B
  The FOLFOX regimen consisted of every 2 weeks cycles for 12 cycles of 2-hour infusions of oxaliplatin at 85 mg/m2 and leucovorin at 400 mg/m2, followed by a bolus infusion of 400-mg/m2 of fluorouracil following by 46-48-hour continuous infusion of 2400-mg/m2 of fluorouracil.
  Celecoxib was dosed at 400 mg orally daily, starting by day 1 of the second treatment of FOLFOX. Celecoxib was administered daily for 3 years from the date of initiation of the first dose or until recurrence of disease or unacceptable toxicity.
  Arm D
  The FOLFOX regimen consisted of every 2 weeks cycles for 6 cycles of 2-hour infusions of oxaliplatin at 85 mg/m2 and leucovorin at 400 mg/m2, followed by a bolus infusion of 400-mg/m2 of fluorouracil following by 46-48-hour continuous infusion of 2400-mg/m2 of fluorouracil.
  Celecoxib was dosed at 400 mg orally daily, starting by day 1 of the second treatment of FOLFOX. Celecoxib was administered daily for 3 years from the date of initiation of the first dose or until recurrence of disease or unacceptable toxicity.
Arm/Group | FOLFOX and Placebo (Arms A +C) | FOLFOX Plus Celecoxib Daily (Arms B + D)
Number analyzed (Participants) | 1261 | 1263
percentage of participants | 73.4 [70.8 to 76.0] | 76.3 [73.8 to 78.8]
Statistical Analysis 1: Comparison: FOLFOX and Placebo (Arms A +C); Test type: Superiority; p = 0.12, Log Rank; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.76 to 1.03]

2. Secondary Outcome: Overall Survival
Description: Overall Survival (DFS) is defined as the time of randomization until documented death from any cause. The endpoint is to compare overall survival of patients with stage III colon cancer randomized to standard chemotherapy only (FOLFOX; Arm A and Arm C) or standard chemotherapy (FOLFOX) with 5 years of celecoxib 400 mg daily (Arm B and Arm D). The percentage of patients who were alive after 3 years are reported here.
Time Frame: up to 3 years from registration
Population: All patients that were randomized and evaluable were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FOLFOX and Placebo (Arms A +C) | FOLFOX Plus Celecoxib Daily (Arms B + D)
Number analyzed (Participants) | 1261 | 1263
percentage of participants | 81.6 [79.4 to 83.9] | 84.3 [82.2 to 86.5]

ADVERSE EVENTS:
Time Frame: Adverse events were collected after every 2-week cycle during treatment (up to 12 cycles or 24 weeks of treatment).
Groups:
- Arm A - FOLFOX and Placebo (12 Treatments); Arm C - 6 Cycles of FOLFOX Plus Placebo Daily: Placebo was dosed at 400 mg orally daily, starting by day 1 of the second treatment of FOLFOX. Placebo was administered daily for 3 years from the date of initiation of the first dose or until recurrence of disease or unacceptable toxicity.
- Arm B - 12 Cycles of FOLFOX Plus Celecoxib Daily; Arm D - 6 Cycles of FOLFOX Plus Celecoxib Daily: Celecoxib was dosed at 400 mg orally daily, starting by day 1 of the second treatment of FOLFOX. Celecoxib was administered daily for 3 years from the date of initiation of the first dose or until recurrence of disease or unacceptable toxicity.
Arm/Group | Arm A - FOLFOX and Placebo (12 Treatments) | Arm B - 12 Cycles of FOLFOX Plus Celecoxib Daily | Arm C - 6 Cycles of FOLFOX Plus Placebo Daily | Arm D - 6 Cycles of FOLFOX Plus Celecoxib Daily
All-Cause Mortality (participants affected / at risk) | 10/615 | 8/647 | 10/646 | 9/618
Serious Adverse Events (participants affected / at risk) | 77/615 | 93/647 | 72/646 | 78/618
Other Adverse Events (participants affected / at risk) | 574/615 | 615/647 | 618/646 | 589/618
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - FOLFOX and Placebo (12 Treatments) (N=615) | Arm B - 12 Cycles of FOLFOX Plus Celecoxib Daily (N=647) | Arm C - 6 Cycles of FOLFOX Plus Placebo Daily (N=646) | Arm D - 6 Cycles of FOLFOX Plus Celecoxib Daily (N=618)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (4)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 (3) | 5 (5) | 6 (6) | 6 (6)
Hemolysis (Blood and lymphatic system disorders) | 3 (4) | 3 (5) | 2 (2) | 7 (7)
Spleen disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asystole (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Cardiac disorder (Cardiac disorders) | 0 (0) | 3 (3) | 3 (3) | 2 (2)
Cardiac pain (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 5 (5) | 11 (11) | 9 (9) | 7 (7)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Optic nerve disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 8 (8)
Anal mucositis (clin exam) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 27 (33) | 33 (35) | 24 (25) | 12 (13)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 3 (4) | 4 (4) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (clin exam) (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (funct/sympt) (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 23 (28) | 22 (24) | 27 (29) | 20 (20)
Pancreatic necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Rectal mucositis (clin exam) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salivary gland disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal mucositis (clin exam) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (2) | 3 (3)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 13 (15) | 10 (12) | 17 (17) | 8 (8)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death NOS (General disorders) | 4 (4) | 0 (0) | 0 (0) | 5 (5)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 41 (47) | 50 (56) | 29 (32) | 30 (30)
Fever (General disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Flu-like symptoms (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gait abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General symptom (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gallbladder fistula (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone infection(unknown ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter related infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalitis infection(unknown ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gallbladder infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Infectious colitis(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious colitis(unknown ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis(unknown ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia(unknown ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sepsis(unknown ANC) (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Soft tissue infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection(unknown ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection(unknown ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urethral infection(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Intestinal stoma obstruction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraoperative breast injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (5)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 11 (13) | 15 (15) | 11 (12) | 11 (11)
Electrocardiogram QTc interval prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 3 (3) | 4 (4) | 4 (4) | 2 (2)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 21 (23) | 26 (30) | 16 (18) | 17 (18)
Platelet count decreased (Investigations) | 25 (27) | 36 (41) | 20 (21) | 8 (9)
Weight gain (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (7) | 1 (1) | 2 (2) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 4 (4) | 8 (9) | 5 (5) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 7 (9) | 7 (7) | 6 (6) | 2 (2)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Serum calcium decreased (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 3 (3) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 5 (6) | 4 (4) | 3 (3) | 4 (4)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (5) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 4 (4) | 0 (0) | 2 (2) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 49 (59) | 54 (64) | 35 (38) | 32 (34)
Radiculitis brachial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bladder pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (3) | 2 (2) | 1 (1) | 2 (2)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 3 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand-and-foot syndrome/reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 13 (13) | 17 (18) | 16 (18) | 16 (21)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Peripheral ischemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 8 (8) | 12 (12) | 8 (17) | 2 (2)
Vascular disorder (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - FOLFOX and Placebo (12 Treatments) (N=615) | Arm B - 12 Cycles of FOLFOX Plus Celecoxib Daily (N=647) | Arm C - 6 Cycles of FOLFOX Plus Placebo Daily (N=646) | Arm D - 6 Cycles of FOLFOX Plus Celecoxib Daily (N=618)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 4 (27) | 4 (15) | 3 (5)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (11) | 12 (14) | 17 (18) | 15 (17)
Hemoglobin decreased (Blood and lymphatic system disorders) | 13 (33) | 23 (51) | 10 (15) | 18 (21)
Hemolysis (Blood and lymphatic system disorders) | 63 (194) | 53 (158) | 49 (102) | 49 (108)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 4 (4) | 6 (10) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 2 (6) | 1 (4) | 0 (0)
Cardiac disorder (Cardiac disorders) | 3 (4) | 2 (2) | 1 (1) | 1 (1)
Cardiac pain (Cardiac disorders) | 0 (0) | 1 (4) | 0 (0) | 2 (2)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 3 (3) | 6 (7) | 4 (4) | 4 (5)
Palpitations (Cardiac disorders) | 0 (0) | 1 (7) | 2 (2) | 2 (4)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 3 (11) | 2 (20) | 1 (7) | 1 (2)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (10) | 1 (1) | 1 (1) | 0 (0)
Endocrine disorder (Endocrine disorders) | 1 (6) | 1 (1) | 2 (2) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 2 (2) | 0 (0) | 3 (9) | 1 (6)
Dry eye syndrome (Eye disorders) | 0 (0) | 1 (3) | 1 (1) | 1 (1)
Eye disorder (Eye disorders) | 1 (1) | 2 (3) | 1 (3) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Optic nerve disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (19) | 0 (0)
Optic nerve edema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 2 (2) | 4 (14) | 4 (10)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (21) | 1 (1) | 1 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 21 (30) | 21 (31) | 19 (26) | 21 (27)
Anal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 2 (2)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colonic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 15 (24) | 11 (21) | 25 (51) | 21 (43)
Diarrhea (Gastrointestinal disorders) | 339 (1107) | 361 (1252) | 353 (922) | 326 (857)
Dry mouth (Gastrointestinal disorders) | 3 (4) | 3 (5) | 2 (8) | 0 (0)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (26) | 7 (9) | 6 (20) | 7 (19)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 2 (2) | 1 (1) | 2 (2)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Esophageal mucositis (clin exam) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Esophageal mucositis (funct/sympt) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (4) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Flatulence (Gastrointestinal disorders) | 3 (9) | 1 (2) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastric mucositis (clin exam) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastric mucositis (funct/sympt) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 5 (9) | 13 (17) | 8 (9) | 9 (12)
Gastritis (Gastrointestinal disorders) | 39 (70) | 40 (64) | 39 (63) | 42 (80)
Gastrointestinal disorder (Gastrointestinal disorders) | 6 (7) | 8 (25) | 3 (4) | 7 (9)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Jejunal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal mucositis (funct/sympt) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (clin exam) (Gastrointestinal disorders) | 6 (6) | 2 (2) | 2 (2) | 5 (5)
Mucositis oral (funct/sympt) (Gastrointestinal disorders) | 12 (16) | 17 (25) | 8 (11) | 9 (10)
Nausea (Gastrointestinal disorders) | 375 (1151) | 395 (1240) | 393 (857) | 360 (844)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (3) | 2 (4) | 2 (3) | 2 (4)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (5) | 4 (5) | 2 (2)
Rectal mucositis (clin exam) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Salivary gland disorder (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 4 (5) | 4 (4) | 3 (4) | 4 (4)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 164 (271) | 167 (283) | 143 (204) | 118 (195)
Chest pain (General disorders) | 1 (3) | 3 (3) | 3 (3) | 0 (0)
Chills (General disorders) | 2 (2) | 1 (1) | 1 (2) | 1 (1)
Edema limbs (General disorders) | 8 (14) | 10 (38) | 9 (15) | 7 (8)
Facial pain (General disorders) | 0 (0) | 1 (1) | 3 (6) | 0 (0)
Fatigue (General disorders) | 471 (2400) | 500 (2649) | 491 (1972) | 456 (1723)
Fever (General disorders) | 5 (5) | 0 (0) | 0 (0) | 3 (3)
Flu-like symptoms (General disorders) | 2 (2) | 0 (0) | 2 (4) | 4 (6)
Gait abnormal (General disorders) | 1 (1) | 2 (8) | 0 (0) | 2 (2)
General symptom (General disorders) | 1 (3) | 2 (3) | 1 (6) | 2 (2)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ill-defined disorder (General disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (3)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Localized edema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pain (General disorders) | 11 (17) | 12 (20) | 14 (22) | 14 (22)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (9)
Cytokine release syndrome (Immune system disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 12 (13) | 7 (8) | 5 (5) | 7 (9)
Immune system disorder (Immune system disorders) | 2 (5) | 0 (0) | 0 (0) | 2 (2)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorectal infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder infection(gr 3/4 ANC) (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Bladder infection(unknown ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone infection(unknown ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis(unknown ANC) (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Catheter related infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis, infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Device related infection(unknown ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endocarditis infective(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gallbladder infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection(gr 0/1/2 ANC) (Infections and infestations) | 4 (4) | 6 (8) | 4 (5) | 4 (4)
Infectious colitis(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infectious colitis(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Infectious meningitis(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney infection(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Laryngitis(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Otitis media(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral nerve infection(unknown ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia(gr 3/4 ANC) (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Pneumonia(unknown ANC) (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Rhinitis infective(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salivary gland infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scrotal infection(unknown ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sepsis(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis(unknown ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinusitis(gr 3/4 ANC) (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 4 (4) | 4 (5) | 3 (7)
Skin infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Skin infection(unknown ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Soft tissue infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Tooth infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory infection(unknown ANC) (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Upper respiratory infectn(gr 0/1/2 ANC) (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection(gr 0/1/2 ANC) (Infections and infestations) | 4 (4) | 3 (3) | 1 (1) | 4 (4)
Urinary tract infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection(unknown ANC) (Infections and infestations) | 0 (0) | 2 (2) | 1 (2) | 3 (3)
Vaginal infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral hepatitis (Infections and infestations) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 4 (5) | 2 (3) | 0 (0)
Wound infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wound infection(gr 3/4 ANC) (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Arterial injury - Extremity-lower (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 4 (5) | 6 (6) | 3 (3) | 1 (1)
Injury to carotid artery (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraop. inj. - Colon (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraop. inj. - Joint (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Intraop. inj. - Small bowel NOS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraop. inj. - Vein-major visceral vein (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraoperative complications (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Intraoperative gastrointestinal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Intraoperative ocular injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Intraoperative urinary injury - Bladder (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 4 (16) | 5 (5) | 9 (19) | 5 (10)
Venous injury - Extremity-lower (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 1 (7) | 0 (0) | 3 (3)
Activated partial throm time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 8 (17) | 10 (29) | 8 (12) | 10 (28)
Alkaline phosphatase increased (Investigations) | 8 (15) | 11 (19) | 1 (1) | 5 (10)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 16 (35) | 14 (39) | 8 (9) | 13 (28)
Blood bilirubin increased (Investigations) | 4 (9) | 4 (6) | 3 (4) | 4 (15)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 76 (256) | 126 (418) | 85 (316) | 100 (306)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (9) | 0 (0)
INR increased (Investigations) | 3 (7) | 8 (21) | 5 (10) | 0 (0)
Laboratory test abnormal (Investigations) | 4 (8) | 2 (3) | 0 (0) | 3 (4)
Leukocyte count decreased (Investigations) | 23 (49) | 27 (43) | 15 (18) | 18 (28)
Lipase increased (Investigations) | 0 (0) | 1 (7) | 2 (4) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (3) | 6 (7) | 4 (4) | 4 (10)
Neutrophil count decreased (Investigations) | 385 (987) | 400 (981) | 303 (564) | 312 (583)
Platelet count decreased (Investigations) | 373 (1552) | 417 (1827) | 332 (828) | 315 (881)
Weight gain (Investigations) | 10 (19) | 12 (33) | 10 (19) | 8 (26)
Weight loss (Investigations) | 9 (10) | 4 (5) | 2 (3) | 4 (8)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 15 (28) | 17 (19) | 8 (9) | 7 (18)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 31 (74) | 47 (100) | 37 (84) | 26 (55)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 17 (24) | 9 (9) | 6 (6)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Obesity (Metabolism and nutrition disorders) | 1 (4) | 2 (12) | 3 (5) | 3 (11)
Serum albumin decreased (Metabolism and nutrition disorders) | 4 (9) | 7 (14) | 5 (5) | 9 (15)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (2) | 3 (10) | 6 (10) | 5 (6)
Serum calcium increased (Metabolism and nutrition disorders) | 3 (5) | 4 (5) | 4 (6) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 4 (4) | 2 (2)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 4 (8) | 3 (5) | 4 (8) | 3 (3)
Serum potassium decreased (Metabolism and nutrition disorders) | 28 (39) | 26 (33) | 23 (28) | 11 (12)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (2) | 3 (4) | 4 (4) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 8 (20) | 6 (14) | 8 (17) | 5 (7)
Serum sodium increased (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Serum triglycerides increased (Metabolism and nutrition disorders) | 2 (2) | 1 (5) | 2 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (17) | 6 (11) | 11 (22) | 5 (8)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (5) | 2 (3) | 1 (1) | 3 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (32) | 12 (36) | 11 (15) | 12 (31)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 4 (7) | 2 (2) | 2 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Joint range motion decr cervical spine (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (6) | 9 (9) | 1 (2) | 4 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 4 (6) | 5 (11) | 5 (7) | 5 (24)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (19) | 4 (11) | 4 (18) | 6 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (9) | 2 (2) | 2 (7) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (31) | 9 (11) | 7 (7) | 6 (12)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3) | 2 (2) | 0 (0)
Accessory nerve disorder (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (6)
Ataxia (Nervous system disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 6 (11) | 10 (12) | 7 (7) | 5 (11)
Dysgeusia (Nervous system disorders) | 6 (11) | 10 (14) | 5 (10) | 5 (8)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 14 (25) | 12 (18) | 8 (14) | 14 (26)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 7 (12) | 7 (7) | 6 (6) | 2 (2)
Memory impairment (Nervous system disorders) | 3 (5) | 2 (4) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 4 (11) | 2 (5) | 2 (2) | 0 (0)
Olfactory nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 3 (6) | 3 (4) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 516 (4338) | 556 (4460) | 501 (2756) | 485 (2662)
Seizure (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (5) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 9 (9) | 9 (10) | 3 (3) | 9 (9)
Syncope vasovagal (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 2 (3) | 2 (3) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 6 (14) | 10 (17) | 10 (18) | 13 (20)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 5 (16) | 5 (8) | 7 (18) | 7 (10)
Insomnia (Psychiatric disorders) | 8 (24) | 10 (19) | 7 (24) | 12 (29)
Irritability (Psychiatric disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bladder hemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Bladder obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (2) | 1 (1)
Hemoglobin urine positive (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
Urinary retention (Renal and urinary disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 1 (1) | 5 (5) | 8 (9) | 2 (3)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 1 (4) | 0 (0) | 1 (1)
Nipple deformity (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (2) | 0 (0) | 5 (13)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4) | 5 (5) | 10 (18)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 10 (12) | 8 (19) | 8 (14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (6) | 2 (3) | 6 (11)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 2 (4) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2) | 2 (2) | 1 (1)
Laryngeal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal mucositis (clin exam) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 3 (4) | 0 (0)
Pharyngeal mucositis (funct/sympt) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (7)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 7 (8) | 3 (3) | 2 (2)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (14) | 9 (15) | 6 (8) | 10 (17)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (4) | 2 (5) | 4 (10)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand-and-foot syndrome/reaction (Skin and subcutaneous tissue disorders) | 8 (13) | 7 (10) | 3 (6) | 5 (6)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (4) | 2 (3) | 0 (0) | 3 (4)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6) | 6 (11) | 2 (2) | 6 (11)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 8 (13) | 1 (1) | 3 (5)
Rash desquamating (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (6) | 4 (8) | 3 (3)
Skin disorder (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (4) | 5 (16) | 6 (8)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (5) | 4 (9) | 0 (0) | 3 (3)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (13) | 1 (8)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 2 (2) | 4 (4)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 2 (2) | 0 (0) | 2 (5) | 1 (1)
Hot flashes (Vascular disorders) | 2 (3) | 5 (16) | 0 (0) | 3 (4)
Hypertension (Vascular disorders) | 216 (1147) | 264 (1474) | 250 (1159) | 252 (1385)
Hypotension (Vascular disorders) | 4 (6) | 4 (6) | 1 (1) | 3 (3)
Peripheral ischemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Phlebitis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 6 (8) | 17 (38) | 16 (24) | 11 (28)
Vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT01150045/Prot_SAP_000.pdf